CLINICAL TRIAL: NCT06843590
Title: A Phase 2, Randomized, Parallel-Group, Double-Blind, Dose-Range-Finding Study to Evaluate the Safety and Efficacy of ALKS 2680 in Subjects With Idiopathic Hypersomnia (Vibrance-3)
Brief Title: A Study to Evaluate the Safety and Effectiveness of ALKS 2680 in Subjects With Idiopathic Hypersomnia
Acronym: Vibrance-3
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALKS 2680-203
Record Dates: First submitted 2025-02-21; First posted 2025-02-25 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Idiopathic Hypersomnia
Keywords: Idiopathic Hypersomnia; IH; sleep; sleep disorder; orexin-2 receptor agonist; excessive daytime sleepiness
MeSH Terms: conditions — Idiopathic Hypersomnia; Sleep Wake Disorders; Disorders of Excessive Somnolence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ALKS 2680, 10 mg (Experimental): Oral tablet containing 10 mg of ALKS 2680 for once daily administration
  Interventions: Drug: ALKS 2680
- ALKS 2680, 14 mg (Experimental): Oral tablet containing 14 mg of ALKS 2680 for once daily administration
  Interventions: Drug: ALKS 2680
- ALKS 2680, 18 mg (Experimental): Oral tablet containing 18 mg of ALKS 2680 for once daily administration
  Interventions: Drug: ALKS 2680
- Placebo (Placebo Comparator): Oral placebo tablet for once daily administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALKS 2680 — Oral tablet containing ALKS 2680 for once daily administration
  Arms: ALKS 2680, 10 mg; ALKS 2680, 14 mg; ALKS 2680, 18 mg
Drug: Placebo — Oral placebo tablet for once daily administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to measure the safety and decrease in daytime sleepiness in subjects with Idiopathic Hypersomnia when taking ALKS 2680 tablets compared with placebo tablets

ELIGIBILITY:
Inclusion Criteria:

* Is willing and able, in the opinion of the Investigator, to understand and comply with protocol requirements, including: lifestyle considerations and restrictions, adherence to contraception guidance, adherence to actigraphy and diary requirements, if receiving treatment for OSA, adherence to primary OSA therapy over the 30 days prior to Visit 1, and throughout the study, including during overnight visits.
* Meets the diagnostic criteria of Idiopathic Hypersomnia according to ICSD-3-TR guidelines, confirmed by the diagnostic evaluations (PSG/MSLT/actigraphy) within the previous 10 years

Exclusion Criteria:

* Has another comorbid sleep disorder or condition that may influence the sleep-wake cycle
* Has a history or presence at Visit 1 of other clinically significant (treated or untreated) illness, disease, abnormality, or surgical procedure that, in the opinion of the Investigator, might compromise subject safety, interfere with any study assessment, or affect the subject's ability to complete the study
* Is currently enrolled in another clinical study or used any investigational drug or device within 30 days prior to Visit 1
* Is currently pregnant, breastfeeding, or is planning to become pregnant during the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Epworth Sleepiness Scale (ESS) from baseline to Week 8 by dose level | Up to 8 weeks

SECONDARY OUTCOMES:
Change in Idiopathic Hypersomnia Severity Scale (IHSS) from baseline to Week 8 by dose level | Up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alkermes, Inc.
Locations (47):
- United States (32):
  - Alkermes Investigator Site, Cullman, Alabama
  - Alkermes Investigator Site, Phoenix, Arizona
  - Alkermes Investigator Site, Little Rock, Arkansas
  - Alkermes Investigator Site, Los Angeles, California
  - Alkermes Investigator Site, Redwood City, California
  - Alkermes Investigator Site, San Francisco, California
  - Alkermes Investigator Site, Colorado Springs, Colorado
  - Alkermes Investigator Site, Brandon, Florida
  - Alkermes Investigator Site, Miami, Florida
  - Alkermes Investigator Site, Winter Park, Florida
  - Alkermes Investigator Site, Atlanta, Georgia
  - Alkermes Investigator Site, Macon, Georgia
  - Alkermes Investigator Site, Stockbridge, Georgia
  - Alkermes Investigator Site, Peoria, Illinois
  - Alkermes Investigator Site, Kansas City, Kansas
  - Alkermes Investigator Site, Lansing, Michigan
  - Alkermes Investigator Site, Lincoln, Nebraska
  - Alkermes Investigator Site, Middletown, New Jersey
  - Alkermes Investigator Site, Denver, North Carolina
  - Alkermes Investigator Site, Huntersville, North Carolina
  - Alkermes Investigator Site, Canton, Ohio
  - Alkermes Investigator Site, Cincinnati, Ohio
  - Alkermes Investigator Site, Cleveland, Ohio
  - Alkermes Investigator Site, Danville, Pennsylvania
  - Alkermes Investigator Site, Philadelphia, Pennsylvania
  - Alkermes Investigator Site, Wyomissing, Pennsylvania
  - Alkermes Investigator Site, Columbia, South Carolina
  - Alkermes Investigator Site, Austin, Texas
  - Alkermes Investigator Site, San Antonio, Texas
  - Alkermes Investigator Site, Sugar Land, Texas
  - Alkermes Investigator Site, Sugarland, Texas
  - Alkermes Investigator Site, Madison, Wisconsin
- Australia (3):
  - Alkermes Investigator Site, Sydney, New South Wales
  - Alkermes Investigator Site, Bedford Park, South Australia
  - Alkermes Investigator Site, Clayton, Victoria
- Belgium (2):
  - Alkermes Investigator Site, Alken
  - Alkermes Investigator Site, Namur
- Alkermes Investigator Site, Prague, Czechia
- France (3):
  - Alkermes Investigator Site, Bordeaux, Gironde
  - Alkermes Investigator Site, Montpellier, Herault
  - Alkermes Investigator Site, Grenoble, Isere
- Italy (3):
  - Alkermes Investigator Site, Bologna
  - Alkermes Investigator Site, Milan
  - Alkermes Investigator Site, Verona
- Alkermes Investigator Site, Zwolle, Netherlands
- Spain (2):
  - Alkermes Investigator Site, Barcelona
  - Alkermes Investigator Site, Madrid

IPD SHARING:
Plan to Share IPD: Undecided